CLINICAL TRIAL: NCT01594177
Title: Dual Blockage With Afatinib and Trastuzumab as Neoadjuvant Treatment for Patients With Locally Advanced or Operable Breast Cancer Receiving Taxane-anthracycline Containing Chemotherapy
Acronym: DAFNE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBG 70; 2011-004704-38 (EudraCT Number)
Record Dates: First submitted 2012-05-03; First posted 2012-05-08 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Unilateral HER2 Positive Breast Cancer
Keywords: DAFNE; GBG 70; GBG; German Breast Group; GBG Forschungs GmbH; Afatinib; neo-adjuvant; HER-2 positive breast cancer; BIBW 2992; 1200.159
MeSH Terms: interventions — Afatinib; Trastuzumab; Paclitaxel; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): Afatinib-Trastuzumab (6 weeks) followed by Afatinib*-Paclitaxel-Trastuzumab (12 weeks) followed by Epirubicin-Cyclophosphamide-Trastuzumab (12 weeks). *only 11 weeks.
  Interventions: Drug: Afatinib; Drug: Trastuzumab; Drug: Paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Afatinib — 20 mg daily for 17 weeks (first two weeks every second day).
Drug: Trastuzumab — First cycle: loading dose 8 mg/kg (day 1 q day 22), thereafter maintenance dose for 9 cycles: 6 mg/kg (day 1 q day 22).
  Other Names: HERCEPTIN
Drug: Paclitaxel — 80 mg/m² i.v. given weekly on day 1 q day 8 for 12 weeks.
Drug: Epirubicin — 90 mg/m² i.v. given on day 1 q day 22 for 4 cycles.
Drug: Cyclophosphamide — 600 mg/m² i.v. given on day 1 q day 22 for 4 cycles.

SUMMARY:
Anthracycline/taxane based combination chemotherapy of at least 18 weeks represents the standard of care in the neoadjuvant setting. In HER2 positive disease trastuzumab is given simultaneously. Neoadjuvant anthracycline-taxane-based chemotherapy given simul-taneously with trastuzumab achieves a pCR rate of approx. 40%. Recent data showed that a double blockade of the HER2 receptor (e.g. trastuzumab + lapatinib; trastuzumab + pertuzumab) given together with a few cycles of chemotherapy can increase the pCR rate by approximately 20%. So far, there is uncertainty, if afatinib (BIBW 2992), an irreversible HER family blocker can lead to an even more complete blockade of the HER2 pathway when given in combination with trastuzumab. The neoadjuvant setting provides the unique opportunity to assess precisely and at short term the effect of systemic treatment by assessing the pCR at surgery. It also allows treating patients with HER2 positive breast cancer before surgery without standard trastuzumab treatment, as, according to current guideline, trastuzumab can also be given sequentially after surgery. The aim of the study is to show that chemotherapy + trastuzumab + afatinib can achieve significant pCR rates.

DETAILED DESCRIPTION:
Primary objectives:

To compare the pathological complete response (pCR = ypT0/is ypN0) rates of neoadjuvant treatment of afatinib in combination with weekly paclitaxel + trastuzumab followed by epirubicin/ cyclophosphamide/ trastuzumab in patients with HER2-positive primary breast cancer.

Secondary objectives:

To determine the rates of ypT0 ypN0; ypT0; ypT0/is; ypN0; and regression grades according to Sinn.

To determine the response rates of the breast tumor and axillary nodes by physical examination and imaging tests (sonography, mammography, or MRI) after 6 weeks of the 2 anti-HER2 agents alone and at surgery.

To determine the breast and axilla conservation rate after treatment. To assess the toxicity and compliance. To correlate skin toxicity and diarrhoea with pCR. To examine and compare pre-specified molecular markers such as EGFR, HER2, HER3, HER4, TGFß, EGF, AREG, HBEGF, BTC, EPIGEN, EREG, NRG1, NRG2, neuroglycan, tomoregulin, NRG4 and NRG3K-RAS, MET, IGF1R, IRS1, PTEN, FGFR1, FGFR2, FGFR3, AXL, RET, and PDGFR; EGFR signature, Ki67, p95HER2, and PI3K mutation before start of afatinib+trastuzumab, before and after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for all study procedures according to local regulatory requirements prior to beginning of specific protocol procedures.
2. Complete baseline documentation must be sent to GBG Forschungs GmbH.
3. Unilateral primary carcinoma of the breast, confirmed histologically by core biopsy. Fine-needle aspiration is not sufficient. Incisional biopsy is not allowed. Tumor lesion in the breast with a sonographical size of ≥ 2 cm in maximum diameter. The lesion has to be measurable in two dimensions, preferably by sonography. In case of inflammatory disease, the extent of inflammation can be used as measurable lesion.
4. Operable or locally advanced or inflammatory breast cancer (cT2 - cT4a-d). In patients with multifocal or multicentric breast cancer, the largest lesion should be measured.
5. Centrally confirmed positive HER2 status detected on core biopsy. HER2-positive is defined as IHC 3+ by a validated test method or FISH/SISH ratio > 2.0. Formalin-fixed, paraffin-embedded (FFPE) breast tissue from core biopsy has therefore to be sent to the Department of Pathology at the Charité, Berlin, prior to regsitration.
6. Centrally confirmed hormone receptor status (ER/PgR).
7. Age ≥ 18 years.
8. Karnofsky Performance status ≥ 80%.
9. Normal cardiac function must be confirmed by ECG and cardiac ultrasound (LVEF or shortening fraction) within 3 months prior to registration. Results must be above 55%.
10. Laboratory requirements:

    Hematology
    * Absolute neutrophil count (ANC) ≥ 2.0 x 109/L and
    * Platelets ≥ 100 x 109/L and
    * Hemoglobin ≥ 10 g/dL (≥ 6.2 mmol/L) Hepatic function
    * Total bilirubin ≤ 1.5x UNL and
    * ASAT (SGOT) and ALAT (SGPT) ≤ 1.5x UNL and
    * Alkaline phosphatase ≤ 2.5x UNL. Renal function
    * Creatinine ≤ 175 µmol/L (2 mg/dL) < 1.5x UNL.
11. Negative pregnancy test (urine or serum) within 14 days prior to registration for all women of childbearing potential.
12. Complete staging work-up within 3 months prior to registration. All patients must have bilateral mammography, breast ultrasound (≤ 21 days), breast MRI (optional), chest X-ray (PA and lateral), abdominal ultrasound or CT scan or MRI, and bone scan done. In case of positive bone scan, bone X-ray is mandatory. Other tests may be performed as clinically indicated.
13. Patients must be available and compliant for treatment and follow-up. Patients registered on this trial must be treated at the participating or at a cooperating centre.

Exclusion Criteria:

1. Bilateral breast cancer.
2. Prior chemotherapy for any malignancy.
3. Prior radiation therapy for breast cancer.
4. Pregnant or lactating patients. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures (barrier methods, intrauterine contraceptive devices, sterilisation) during study treatment.
5. Inadequate general condition (not fit for anthracycline-taxane based chemotherapy) as per investigator´s assessment.
6. Previous malignant disease with a disease-free period of less than 5 years (except CIS of the cervix and non-melanomatous skin cancer).
7. Known or pre-existing interstitial lung disease.
8. Known or suspected congestive heart failure (NYHA > I) or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, uncontrolled or poorly controlled arterial hypertension (i.e. BP > 160/90 mm Hg under treatment with two antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease.
9. History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent.
10. Chronic-inflammatory bowel diseases.
11. Pre-existing motor or sensory neuropathy of a severity grade ≥ 2 by NCI-CTCAE criteria.
12. No evidence or history of infection (including hepatitis B, C or HIV).
13. Known hypersensitivity reaction to one of the investigational compounds or incorporated substances used in this protocol.
14. Definite contraindications for the use of corticosteroids except inhalative corticoids.
15. Concurrent treatment with:

    * chronic corticosteroids unless initiated > 6 months prior to study entry and at low dose (≤ 10 mg methylprednisolone or equivalent).
    * sex hormones. Prior treatment must be stopped before study entry.
    * other experimental drugs or any other anti-cancer therapy.
16. Participation in another clinical trial with any investigational, not marketed drug within 30 days prior to study entry.
17. Male patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response | 30 weeks
  To compare the pathological complete response (pCR = ypT0/is ypN0) rates of neoadjuvant treatment of afatinib in combination with weekly paclitaxel + trastuzumab followed by epirubicin/ cyclophosphamide/ trastuzumab in patients with HER2-positive primary breast cancer.

SECONDARY OUTCOMES:
Pathological Complete Response | 30 weeks
  To determine the rates of ypT0 ypN0; ypT0; ypT0/is; ypN0; and regression grades according to Sinn.
Response Rate by Physical Examination and Imaging Tests | 30 weeks
  To determine the response rates of the breast tumor and axillary nodes by physical examination and imaging tests (sonography, mammography, or MRI) after 6 weeks of the 2 anti-HER2 agents alone and at surgery.
Conservation Rate | 30 weeks
  To determine the breast and axilla conservation rate after treatment.
Number of Participants with (Serious) Adverse Events as a Measure of Safety and Tolerability | 30 weeks
  Analysis of number and grading of (serious) adverse events during the different treatment phases.
Number of Participants with Skin Toxicity and Diarrhea as (Serious) Adverse Events as a Measure of Safety and Tolerability and Pathological Complete Response | 30 weeks
  Analysis of number and grading of skin toxicity and diarrhea as (serious) adverse events in correlation with pCR.
Translational Research | 30 weeks
  To examine and compare pre-specified molecular markers such as EGFR, HER2, HER3, HER4, TGFß, EGF, AREG, HBEGF, BTC, EPIGEN, EREG, NRG1, NRG2, neuroglycan, tomoregulin, NRG4 and NRG3K-RAS, MET, IGF1R, IRS1, PTEN, FGFR1, FGFR2, FGFR3, AXL, RET, and PDGFR; EGFR signature, Ki67, p95HER2, and PI3K mutation before start of afatinib+trastuzumab, before and after chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Claus A Hanusch, MD, PhD, Principal Investigator — Rotkreuzklinikum München, 80634 München, Rotkreuzplatz 8
Locations (1):
- Rotkreuzklinikum München, München, Germany